CLINICAL TRIAL: NCT07146295
Title: Implementation of Fluorescent Imaging Using Indocyanine Green to Identify Sentinel Lymph Nodes During Surgery for Breast Cancer
Brief Title: Implementation of Indocyanine Green to Identify Sentinel Lymph Nodes During Surgery for Breast Cancer
Acronym: INFINITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isabelle Henskens (Other)
Collaborators: Canisius-Wilhelmina Hospital (Other); Spaarne Gasthuis (Other); Noordwest Ziekenhuisgroep (Other); Alrijne Hospital (Other); Dijklander Ziekenhuis (Other); Ziekenhuisgroep Twente (Other); Diakonessenhuis, Utrecht (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor-Investigator, Isabelle Henskens, Coordinating investigator, St. Antonius Hospital
Organization: St. Antonius Hospital (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: NL87551.100.24; 10390172310041 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2025-08-08; First posted 2025-08-28 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Sentinel Lymph Node Biopsy (SLNB); Sentinel Lymph Node Detection; Sentinel Lymph Node; Lymphatic Metastasis; Fluorescence Imaging; Indocyanine Green (ICG); Radioisotopes; Lymph Node Mapping
Keywords: Breast cancer; Sentinel lymph node biopsy; Lymphatic metastasis; Indocyanine green; Techetium nanocolloïd; Fluorescence imaging; Surgical oncology; Lymph node mapping; Implementation; Radioisotope
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis | interventions — Technetium; Technetium-99; Indocyanine Green; Optical Imaging; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Intervention Model Description: This is a stepped-wedge cluster trial in which participating hospitals (clusters) are selected to represent different regions, settings, and sizes. The order in which hospitals transition is based on site readiness and in consultation with the participating centers. All hospitals begin with the current standard of care using radioisotope technetium-labeled (99mTc)-nanocolloid for sentinel lymph node biopsy (SLNB). At fixed intervals, clusters move to a transition phase using both 99mTc and indocyanine green (ICG), and then to ICG only. This sequential rollout creates an iterative learning cycle, allowing evaluation of the implementation process and refinements between phases. The total study duration is 18 months, with a fixed 6-month transition phase per cluster.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-implementation (99mTc only) (Active Comparator): Participants undergo sentinel lymph node biopsy (SLNB) using the current standard of care: injection of radioisotope technetium-labeled (99mTc)-nanocolloid and preoperative lymphoscintigraphy, followed by radio-guided surgery with a gamma-detection probe.
  Interventions: Drug: Technetium (99mTc); Drug: Indocyanine Green; Procedure: Sentinel lymph node biopsy
- Transition phase (99mTc + ICG) (Experimental): Participants receive preoperative injection of radioisotope technetium-labeled (99mTc)-nanocolloid and preoperative lymphoscintigraphy (without marking the location on the skin). Surgeons are blinded to preoperative lymphoscintigraphy results. After induction of general anesthesia, indocyanine green (ICG) is injected periareolar. Surgery is primarily guided by ICG fluorescence imaging to identify and remove the sentinel lymph node(s). Excised lymph nodes are then checked for 99mTc activity using a gamma-detection probe as a control. This phase is designed to allow surgeons to gain experience with the ICG technique while maintaining safety through parallel use of the established 99mTc method.
  Interventions: Drug: Indocyanine Green; Procedure: Sentinel lymph node biopsy
- Post-implementation (ICG only) (Active Comparator): Participants undergo SLNB using ICG only. ICG is injected periareolar after induction of general anesthesia and visualized intraoperatively with a fluorescence camera to guide excision of the sentinel lymph node(s).
  Interventions: Drug: Technetium (99mTc); Procedure: Sentinel lymph node biopsy

INTERVENTIONS:
Drug: Technetium (99mTc) — A radiopharmaceutical tracer consisting of technetium-99m (99mTc)-labelled nanocolloid used for sentinel lymph node mapping. In this study, 99mTc-nanocolloid is administered via periareolar injection with an activity of 40 MBq for the one-day protocol or 100 MBq for the two-day protocol, according to local hospital practice. Injection is performed either on the day of surgery or the afternoon before surgery. Preoperative lymphoscintigraphy is carried out to visualize lymphatic drainage. During surgery, a gamma-detection probe is used to locate and remove the sentinel lymph node(s) identified by 99mTc uptake.
  Other Names: 99mTc; Technetium-99m labelled nanocolloid; Technetium-99; Technetium-99m; Tc99
  Arms: Post-implementation (ICG only); Pre-implementation (99mTc only)
Drug: Indocyanine Green — Indocyanine Green (ICG) is a fluorescent dye used for intraoperative sentinel lymph node mapping. In this study, a total dose of 5 mg (2 mL) of ICG is administered via periareolar injection after induction of general anesthesia and prior to axillary incision. During surgery, near-infrared fluorescence imaging is used to visualize lymphatic drainage and identify the sentinel lymph node(s). The identified node(s) are surgically removed under fluorescence guidance. In the transition phase, fluorescence findings are cross-checked against 99mTc uptake to ensure accuracy and safety.
  Other Names: ICG; fluorescence imaging
  Arms: Pre-implementation (99mTc only); Transition phase (99mTc + ICG)
Procedure: Sentinel lymph node biopsy — Sentinel lymph node biopsy (SLNB) is a surgical procedure used to identify and remove the first lymph node(s) that drain lymph from a tumor area. In this study, SLNB is performed through a small axillary incision after mapping the sentinel lymph node(s) using either radioisotope technetium-labeled (99mTc)-nanocolloid, indocyanine green (ICG) fluorescence imaging, or a combination of both. The identified lymph node(s) are excised and sent for pathological examination to determine the presence of cancer cells. The procedure is carried out under general anesthesia as part of breast cancer surgery.
  Other Names: Sentinel lymph node mapping; SLNB; SLN procedure; Sentinel lymph node procedure

SUMMARY:
The goal of this clinical trial is to learn how to successfully introduce a new method for finding the sentinel lymph node during breast cancer surgery into routine hospital care. The method uses a dye called indocyanine green (ICG) and a special camera to see the lymph node. The sentinel lymph node is the first lymph node that cancer is likely to spread to.

In the Netherlands, about 1 in 7 women develops breast cancer. Finding out whether cancer has spread to the lymph nodes is important for planning treatment and predicting outcomes. The current standard method for sentinel lymph node biopsy (SLNB) uses a radioactive tracer called radioisotope technetium-labeled (99mTc)-nanocolloid. While accurate, this method has several drawbacks: it exposes patients to radioactivity, requires an extra hospital visit or travel to another hospital due to limited nuclear medicine facilities, and is not sustainable. Surgeries using 99mTc can only take place on certain days due to logistical issues, and the signal from 99mTc can be disturbed by the tumor marker placed in the breast.

ICG works as well as 99mTc for SLNB and offers several advantages: it is given during surgery (no extra visit needed), produces no radiation, and reduces costs. However, it is still not widely used in the Netherlands because hospitals may not be familiar with it or unsure how to make the switch.

This study will introduce ICG step-by-step in several Dutch hospitals and evaluate how to make the change as smooth and effective as possible. It will take place in three stages: I) SLNB with 99mTc only (current practice); II) SLNB with both 99mTc and ICG (transition phase); III) SLNB with ICG only (full implementation).

All study procedures take place during planned surgery, with no extra hospital visits. After surgery, participants will receive a short questionnaire (10-15 minutes) to share their experiences with the procedure. Their feedback, combined with input from healthcare providers, will help researchers develop a uniform medical protocol, an implementation guide, and educational materials for surgeons and surgical trainees.

The aim is to make ICG widely available across the Netherlands, ensuring that care is less burdensome, more sustainable, and more cost-effective, while keeping treatment accessible in local hospitals.

DETAILED DESCRIPTION:
Background:

Breast cancer affects one in seven women. Detecting lymph node metastases via the sentinel lymph node biopsy (SLNB) is crucial for prognosis and treatment. The gold standard is radio-guided surgery using the radioisotope technetium-labeled (99mTc)-nanocolloid, which requires preoperative injection and lymphoscintigraphy. However, the use of 99mTc poses significant burdens on patients, as it requires additional hospital visits or travel to another hospital due to the limited availability of nuclear medicine facilities. The use of 99mTc also creates logistical challenges and lacks sustainability. A recently proven, equally effective and safe alternative method is peroperative real-time fluorescence imaging using Indocyanine Green (ICG). ICG offers many advantages over 99mTc for patients, healthcare providers, and society. Yet, the use of ICG for SLNB remains limited, as hospitals face challenges due to uncertainty in transitioning and limited familiarity with recent findings. Implementation guidance is imperative for effective adoption, to avert further practice variation and to ensure patients benefit from this evidence-based alternative method.

Objectives:

The INFINITE trial aims to successfully implement ICG-fluorescence for identifying the sentinel lymph node by guiding the implementation process using the Effective Implementation of Change model developed by Grol and Wensing, identifying and understanding the factors influencing implementation outcomes through the Consolidated Framework for Implementation Research, evaluating the outcomes of implementation efforts using a mixed-methods approach and the outcomes framework proposed by Proctor et al., and creating conditions for nationwide implementation. Secondary aims are to develop a uniform medical protocol for the use of ICG for SLNB, to develop an implementation guide that aligns with current practice, to prepare educational materials for surgeons and modules for the curriculum of surgical residents (CASH), to produce patient information materials and organize interactive meetings for surgical healthcare providers and their teams, to further substantiate the effectiveness, safety, and cost-effectiveness of ICG, to increase support and a sense of urgency for ICG implementation by organizing informational sessions during annual conferences of the relevant scientific associations, and to facilitate nationwide scale-up by incorporating ICG into SLNB guidelines.

Study Design:

ICG will be implemented in seven strategically chosen Dutch hospitals during the INFINITE trial. These hospitals have been selected to represent different areas, settings, and sizes, ensuring broad applicability and support for subsequent nationwide implementation. The INFINITE trial is a multicenter hybrid effectiveness-implementation study using a stepped-wedge cluster trial design across three phases: Phase I, pre-implementation (99mTc only); Phase II, transition period (99mTc and ICG); and Phase III, post-implementation (ICG only). Based on site readiness and in consultation with the participating centers, three clusters will be formed, each consisting of two or three hospitals. Clusters will transition to the next phase at fixed intervals, creating an iterative learning cycle. This approach allows for regular evaluations of the implementation strategies, processes, and products, including the protocol, implementation guide, educational materials, and patient information. Process evaluations will inform adjustments using the ERIC-CFIR matching tool, ensuring rapid integration of lessons learned to enhance implementation in the next cluster.

Intervention:

In Phase I, pre-implementation, SLNB is performed using standard care with 99mTc injection and lymphoscintigraphy the day or morning before surgery, followed by radio-guided surgery with a gamma-detection probe. In Phase II, the transition period, SLNB is performed using both ICG and 99mTc. Patients receive 99mTc injection and lymphoscintigraphy before surgery, with the surgeon blinded to the imaging results. During surgery, after induction of general anesthesia and before axillary incision, 5 mg (2 ml) ICG is injected periareolarly, and SLNB is performed using fluorescence imaging. After excision of the sentinel lymph node(s), the standard gamma probe is used to test the excised nodes and the axilla for 99mTc activity, and the axilla is also explored by direct visualization and palpation. In Phase III, post-implementation, SLNB is performed using ICG as the sole tracer, with the same dosage and injection method, and the sentinel lymph node is visualized using fluorescence imaging and excised.

Outcomes:

Study endpoints are categorized into actual and anticipated implementation outcomes, client outcomes, and service outcomes. The primary endpoint is adoption, defined as the proportion of SLNB procedures conducted with ICG only, 99mTc only, or both during Phase III, compared to the total SLNBs in that phase, measured using screening logs and hospital records. All other outcomes are secondary. Fidelity, another actual implementation outcome, is measured through an intraoperative survey. Anticipated implementation outcomes such as appropriateness, feasibility, and acceptability are evaluated via a healthcare provider survey during Phase III. Client outcomes include patient satisfaction assessed through a post-procedure survey. Service outcomes encompass effectiveness, safety, cost-effectiveness, and the impact on necessary personnel, evaluated using perioperative and hospital administration data.

Risks and Burden:

Patients who consent will not experience any extra burden from ICG-fluorescence. ICG will be administered under general anesthesia, so patients will not experience additional discomfort, site visits, or procedures. ICG is non-ionizing and has very few reported complications or adverse events. Considering a maximum of two additional nodes sampled, the preferred anatomical location of these nodes, and the clinical experience with additional lymph node sampling, no increase in surgical morbidity is expected. Patients may benefit from the intervention as ICG can increase sentinel lymph node identification rates and eliminate the need for a preoperative visit to the Nuclear Medicine department for 99mTc injection. Completion of the patient satisfaction questionnaire will take approximately 10 to 15 minutes. Both risks and burden are therefore considered negligible.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old.
* DCIS or invasive breast cancer, confirmed by biopsy
* Clinically node-negative, confirmed by preoperative axillary ultrasound
* Indication for breast cancer surgery with SLN procedure via axillar incision

Exclusion Criteria:

* Combined MARI procedure
* Known allergy for Indocyanine Green (ICG), intravenous contrast or iodine
* History of axillary lymph node dissection
* Hyperthyroidism or thyroid cancer
* Pregnancy or breast-feeding
* No written informed consent according to ICH/GCP and national regulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1760 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Adoption of ICG for sentinel lymph node biopsy (SLNB) | During Phase III, the post-implementation period, which is the final 9 months for hospitals in cluster 1, final 6 months for cluster 2, and final 3 months for cluster 3, within the 18-month trial.
  Proportion of SLNB procedures performed using indocyanine green (ICG) only, compared to the total number of SLNB procedures perfomed, using any tracer, on the target population in the observational cohort of phase III. Adoption will be assessed using hospital administrative data, with cross-checking against the prospective screening and inclusion log.

SECONDARY OUTCOMES:
Fidelity of ICG-fluorescence implementation | Phase III; intraoperative survey completed immediately after each SLNB procedure.
  Degree to which the sentinel lymph node biopsy (SLNB) procedure using indocyanine green (ICG) fluorescence is performed as intended according to the developed protocol. Measured by identifying deviations from the established protocol through an intraoperative survey completed by the operating surgeon.
Appropriateness of ICG-fluorescence | A questionnaire is administered to healthcare providers in each participating hospital during the 3rd month of Phase III, corresponding to month 12 for cluster 1, month 15 for cluster 2, and month 18 for cluster 3.
  Perceived fit, relevance, and compatibility of ICG use for SLNB within the clinical workflow of participating hospitals. Measured at the provider level using a structured questionnaire assessing perceived clinical usefulness, integration into existing practice, and alignment with patient care goals. The questionnaire uses a 5-point Likert scale with a minimum score of 1 and a maximum score of 5. Higher scores indicate better appropriateness.
Feasibility of ICG-fluorescence implementation | A questionnaire is administered to healthcare providers in each participating hospital during the 3rd month of Phase III, corresponding to month 12 for cluster 1, month 15 for cluster 2, and month 18 for cluster 3.
  Extent to which ICG use for SLNB can be successfully carried out within the resources, organizational structure, and time constraints of each participating hospital. Measured via healthcare provider questionnaire assessing practical implementation challenges. The questionnaire uses a 5-point Likert scale with a minimum score of 1 and a maximum score of 5. Higher scores indicate better feasibility.
Acceptability of ICG-fluorescence implementation | A questionnaire is administered to healthcare providers in each participating hospital during the 3rd month of Phase III, corresponding to month 12 for cluster 1, month 15 for cluster 2, and month 18 for cluster 3.
  Satisfaction and acceptance of ICG use for SLNB among healthcare providers. Measured through structured provider questionnaires evaluating perceived benefits, challenges, and willingness to continue using ICG. The questionnaire uses a 5-point Likert scale with a minimum score of 1 and a maximum score of 5. Higher scores indicate better acceptability.
Patient satisfaction with SLNB procedure | Questionnaire administered within 1 week after surgery during all phases of the trial (from study start up to 18 months).
  Satisfaction of participants undergoing SLNB using ICG, 99mTc, or both. Measured at the patient level using phase-specific structured questionnaires administered after surgery. The questionnaires assess understanding of the procedure, clarity of information, burden of additional appointments, pain or discomfort, cosmetic effects (e.g. temporary skin discoloration), and perceived exposure to radioactivity where applicable. Most items are scored on a 5-point Likert scale, where higher scores may reflect either greater burden or greater satisfaction depending on the item. The overall satisfaction item is scored on a 5-point Likert scale with a minimum score of 1 and a maximum score of 5, where higher scores indicate greater satisfaction. In addition, tracer preference is assessed on a 5-point Likert scale ranging from strong preference for ICG to strong preference for Technetium. An open-ended question captures reasons for tracer preference.
Total number of lymph nodes removed, SLNs, and non-SLNs | Intraoperative survey completed immediately after each SLNB procedure across all study phases (from study start up to 18 months).
  The total number of lymph nodes excised during SLNB and sent for pathological examination, including the total number of SLNs, the total number of non-SLNs, and the mean number of nodes excised per SLNB.
Per-node detection of SLNs by tracer | Intraoperative survey completed immediately after each SLNB procedure across all study phases (from study start up to 18 months).
  Count and proportion of excised SLNs identified intraoperatively by ICG, 99mTc, both, or neither. Non-SLNs are excluded. This represents the per-node detection rate.
Tracer Concordance of SLNs | Intraoperative survey completed immediately after each SLNB procedure during Phase II only.
  Proportion of excised SLNs detected by both ICG and 99mTc compared to those detected by only one tracer. Reported as the percentage of SLNs fluorescent but not 99mTc-positive and vice versa. Non-SLNs are excluded.
Per-case identification rate of SLNs by tracer | Intraoperative survey completed immediately after each SLNB procedure across all study phases (from study start up to 18 months).
  Proportion of SLNB procedures in which at least one SLN is identified by the assigned tracer. Reported separately for: Phase I (Tc-99m only), Phase III (ICG only), and Phase II descriptively (tracer-specific rates for Tc-99m and ICG, and combined). This represents the per-case identification rate, including cases of mapping failure.
Paired per-case detection rate of SLNs by ICG versus 99mTc | Intraoperative survey completed immediately after each SLNB procedure during Phase II only.
  Paired comparison in which both ICG and 99mTc are used within the same patient. Proportion of SLNB procedures in which at least one SLN is identified by ICG versus 99mTc, reported as a within-patient comparison.
Detection time to first, second and/or third (sentinel) lymph node | Intraoperative survey completed immediately after each SLNB procedure across all study phases (from study start up to 18 months).
  Minutes from axillary incision to excision of the first, second and/or third (sentinel node); recorded intraoperatively.
Total SLNB procedure duration | Intraoperative survey completed immediately after each SLNB procedure across all study phases (from study start up to 18 months).
  Minutes from axillary skin incision to closure of the axillary wound.
Pathology of SLNs | Data collected from the pathology report within 2-3 weeks after surgery, across all study phases (from study start up to 18 months).
  Pathology results of excised SLNs, summarized per node and per patient: number examined at pathology and number classified as benign, with isolated tumor cells, micrometastasis, or macrometastasis. Analyses will be stratified by tracer and study phase (Phase I: 99mTc; Phase II: dual tracer; Phase III: ICG).
Safety of ICG-fluorescence for SLNB | Events are systematically recorded using a standardized postoperative case report form in REDCap, completed within 3 to 4 weeks after surgery in all study phases (from study start up to 18 months).
  Incidence of perioperative (serious) adverse events potentially related to the use of ICG-fluorescence during SLNB.
Direct in-hospital per-patient costs per SLNB ICG compared to 99mTc | Conducted in parallel with the current study. The cost overview is based on cost drivers associated with each surgical pathway, as identified from the literature and clinical experience.
  This outcome measures the direct in-hospital costs per patient for SLNB comparing the two surgical pathways of ICG and 99mTc-guided SLNB. The analysis includes costs related to equipment, consumables, diagnostics, histopathology, and outpatient care, covering the period from the day before surgery until hospital discharge. Sources for cost determination include Dutch Costing Guidelines (DCG), manufacturer price lists, and the hospital's financial ledger. Costs are calculated by multiplying unit costs with actual resource use.
National budget impact of ICG-fluorescence implementation | Conducted in parallel with the current study. The BIA covers the period of 2025-2029.
  A budget impact analysis from the provider's perspective will be performed using the tool developed by ZonMw to evaluate annual and cumulative five-year national savings and assess the economic impact of phased implementation of ICG on the Dutch healthcare system across 70 institutions within the Dutch healthcare system.
Patient-level costs for SLNB using 99mTc or ICG-fluorescence | Patient survey administered within 1 week after surgery during Phase I (99mTc) and Phase III (ICG).
  Participant-reported travel distance, sick-leave duration, and childcare hours converted into monetary values using national unit-cost references.

CONTACTS AND LOCATIONS:
Overall Officials: Annemiek Doeksen, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (7):
- Netherlands (7):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Ziekenhuisgroep Twente, Hengelo
  - Spaarne Gasthuis, Hoofddorp
  - Dijklander Ziekenhuis, Hoorn
  - Alrijne Hospital, Leiden
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Diakonessenhuis, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided
At present, there is no final decision regarding sharing of individual participant data (IPD). Data sharing will depend on ethical approval, participant consent, and compliance with applicable privacy regulations. If IPD sharing is pursued, only de-identified datasets relevant to the research question will be made available upon reasonable request to qualified researchers, under a data use agreement ensuring confidentiality and scientific integrity